CLINICAL TRIAL: NCT05971303
Title: Examining the Impact of Culturally and Linguistically Diverse Backgrounds on Patient Care and Experiences in Women With Gynecologic Malignancies (iCALD-2): A Questionnaire Study
Brief Title: Impact of Cultural and Linguistic Backgrounds on Patient Care and Experience of Women With Gynecologic Malignancies
Acronym: iCALD-2
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 20-5744
Record Dates: First submitted 2021-05-31; First posted 2023-08-02 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Gynecologic Cancer
Keywords: Visible minority; Linguistic Diversity; Cultural Diversity; Socioeconomic Status; Health Literacy; Patient Care; Patient Experience
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient Questionnaire: Eligible patients will be matched to complete questionnaires in their specified preferred language. Questionnaire patient responses will also be in the patient's identified preferred language, and will be translated into English for study analysis by UHN Interpretation and Translation Services. The questionnaire will comprise of sections in multiple choice and free-text format, administered in an outpatient setting. Question domains will encompass patient demographics, comprehension of diagnosis and treatment, clinical trials, palliative care and overall experiences in the clinic from the perspective of a CALD oncology patient, including identification of any barriers to optimal care.
  Interventions: Other: Questionnaire
- Interpreter Questionnaire: Interpreters will be screened by investigators and approached for their willingness to complete the questionnaires. The questionnaire will comprise of several sections in rating scale and free-text format. Questionnaires will be delivered in English only. Question domains will encompass demographics, professional background, and overall experiences in the clinic setting from the perspective of a professional team member caring for the oncology patient with CALD background, including identification of any barriers to optimal care.
  Interventions: Other: Questionnaire
- Cancer Care Professional Questionnaire: Cancer Care Professionals will be screened by investigators and approached for their willingness to complete the questionnaires. The questionnaire will comprise of several sections in rating scale and free-text format. Questionnaires will be delivered in English only. Question domains will encompass demographics, professional background, and overall experiences in the clinic setting from the perspective of a professional team member caring for the oncology patient with CALD background, including identification of any barriers to optimal care.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires will be given to patients, interpreters and cancer car professionals with aims of delineating the attitudes and experiences of patients, interpreters and cancer care professionals involved in the care of oncology patients with gynecologic malignancies

SUMMARY:
Purpose of this study to delineate the attitudes and experiences of patients, interpreters and cancer care professionals involved in the care of oncology patients with gynecologic malignancies with cultural and linguistic diversity backgrounds, in addition to highlighting any barriers to optimal patient care through questionnaires.

DETAILED DESCRIPTION:
Approximately 45% of Toronto residents have a mother tongue other than English, and over a quarter of people speak a language other than English most often at home, with over 180 different languages and dialects spoken throughout the Greater Toronto Area. Additionally, based on the census data from 2016 there also appears to be an unbalanced distribution between minority background and socioeconomic status, with lower income neighborhoods being primarily occupied by visible minority populations, which has been associated with lower socioeconomic status and poorer health literacy, and potentially correlates with healthcare service utilization overall and worse clinical outcomes.

Although linguistically diverse patients in predominantly Caucasian societies is a common phenomenon, it is relatively poorly studied across the globe, although some reports have demonstrated a tendency towards longer inpatient lengths of stay and higher readmission rates. In particular, one retrospective cohort study at two hospital affiliated with the University of Toronto, Canada, found that in over 9000 patients who presented to the emergency room or were admitted, culturally and linguistically diverse (CALD) patients had higher rates of re-presentations and readmissions if their underlying pathology was a chronic condition (chronic airways disease or cardiac failure) due to the complex care pathways involved upon discharge. This is highly relevant to the oncology patient, as consultations are time-restricted and management algorithms are highly complex and involve multiple parallel communication pathways, which carries a higher risk of misinterpretation when coupled with a background where English is not the patient's primary spoken language.

The use of a professional interpreter in medical consultations, defined by the Ontario Council on Community Interpreting (OCCI) as a "fluently bilingual individual with appropriate training and experience who is able to interpret with consistency and accuracy and who adheres to the Standards of Practice and Ethical Principles," has been shown to reduce significantly medical communication errors as compared with ad-hoc family members, improve duration of hospitalization, reduce readmission rates and improve patient satisfaction.

Caring for patients who come from CALD backgrounds poses a unique set of challenges not only from the perspective of the patient, but also for the treating physicians and team of health professionals, including those employed by interpretation services.

The iCALD-2 protocol aims to investigate barriers affecting CALD patient care using a questionnaire approach. Collectively with the iCALD retrospective study, this protocol looks to establish a baseline from which interventional studies surrounding CALD patients and interpretive services can be launched in the future, with a view to potential expansion across other tumour site clinics .

ELIGIBILITY:
Patient Questionnaires:

Inclusion Criteria:

* Patients who have received anti-cancer treatment and continue to be followed up at Princess Margaret Cancer Centre for a confirmed gynecologic malignancy.
* Patients who have received anti-cancer treatment and continue to be followed up at Princess Margaret Cancer Centre for a confirmed gynecologic malignancy.
* Patients self-identify their preferred spoken and/or written language to be a language other than English.
* The patient's self-identified preferred language is one of the languages in which the questionnaire has been translated.
* Patients must be >18 years old.
* Patients must be willing and able to complete a questionnaire (in their primary written language) as a patient in the oncology clinic independently.
* Life expectancy greater than 3 months.
* Patients must be able to provide written consent with the assistance of a professional interpreter.

Exclusion Criteria:

• Patients must be willing and able to complete the questionnaire independently without the assistance of others.

Interpreter Questionnaires:

Inclusion Criteria:

* Interpreters must have provided medical interpretive services in a professional context for at least 3 months.
* Interpreters must be willing and able to complete a questionnaire detailing their demographics and experiences working as a medical interpreter.
* Interpreters must have experience providing medical interpretive services in an oncology or palliative care setting.

Cancer Care Professional Questionnaires:

Inclusion Criteria:

* Physicians must be staff physicians, fellows, physician assistants, or residents in oncology or palliative care, who are experienced in providing medical care to CALD oncology patients in the context of gynecology or palliative care clinics.
* Other cancer care professionals eligible to participate include but are not limited to nurses, clinical research coordinators, social workers, dietitians, pharmacists, psychologists, and administrative staff.
* Cancer care professionals (except for administrative staff) must have had at least 3 months experience providing clinical care in an oncology or palliative care setting, and must have experience delivering care to CALD patients in this context.
* Administrative staff must have at least 3 months experience working in the context of an oncology or palliative care clinic, and must have regular in-person or by phone patient contact. They must also have experience interacting with patients or carers from CALD backgrounds in an oncology/palliative care setting.
* Cancer care professionals must be willing and able to complete a questionnaire independently detailing their demographics and experiences in treating CALD oncology or palliative care patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients, interpreters and cancer care professionals involved in the care of oncology patients with gynecologic malignancies with culturally and linguistically diverse (CALD) backgrounds.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To describe culturally and linguistically diverse (CALD) patient experiences and attitudes in the clinic setting concerning interpretation services, in addition to barriers to providing care and self-management supports. | 4 to 6 weeks
  •Eligible patients will be matched to complete questionnaires in their specified preferred language. Question domains will encompass patient demographics, comprehension of diagnosis and treatment, clinical trials, palliative care and overall experiences in the clinic from the perspective of a CALD oncology patient, including identification of any barriers to optimal care.
To describe training processes and challenges faced by interpreters when providing services to oncology and palliative care CALD patients. | 4 to 6 weeks
  Questionnaires will be anonymous and delivered in English only. Question domains will encompass demographics, professional background, and overall experiences in the clinic setting from the perspective of a professional team member caring for the oncology patient with CALD background, including identification of any barriers to optimal care.
To describe challenges faced by treating physicians and allied health professionals when providing care to CALD patients in oncology or palliative care clinic settings. | 4 to 6 weeks
  Questionnaires will be anonymous and delivered in English only. Question domains will encompass demographics, professional background, and overall experiences in the clinic setting from the perspective of a professional team member caring for the oncology patient with CALD background, including identification of any barriers to optimal care.

SECONDARY OUTCOMES:
To characterize the demographics of the CALD population in the gynecology clinic with regards to visible minority populations and self-reported preferred first languages. | 4 to 6 weeks
  Frequencies and proportions for the answers of multiple-choice questions in Oncology clinic experiences, Clinical trials and Palliative care clinic sections of Patient Questionnaire will be calculated and reported.
To compare patient distress levels between different ethnic minorities using Distress Assessment and Response Tool (DART) data from iCALD (UHN Research Ethics Board #20-5032) | 4 to 6 weeks
  Patients answer specific questions about physical, emotional and practical challenges that impact with their ability to engage in their cancer care.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L'Heureux, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada